CLINICAL TRIAL: NCT06301555
Title: Game-Based Digital Intervention for Relieving Depression and Anxiety Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: db2023
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blank Control (No Intervention): No intervention
- RL Algorithm Intervention (Experimental)
  Interventions: Behavioral: Reinforcement learning algorithm powered cognitive and behavioral intervention
- No Algorithm Active Control (Active Comparator)
  Interventions: Behavioral: cognitive and behavioral intervention

INTERVENTIONS:
Behavioral: Reinforcement learning algorithm powered cognitive and behavioral intervention — Reinforcement learning algorithm powered cognitive and behavioral intervention
  Arms: RL Algorithm Intervention
Behavioral: cognitive and behavioral intervention — cognitive and behavioral intervention
  Arms: No Algorithm Active Control

SUMMARY:
Objective: To collect preliminary data and assess the preliminary effectiveness of a game-based digital therapeutics (DTx) intervention for individuals with symptoms of anxiety and depression, and to investigate whether reinforcement learning (RL) can personalize the intervention and enhance effectiveness. Design: Randomized controlled trial with three arms. Setting: Internet-based recruitment and delivery of the intervention. Participants: 223 individuals with symptoms of anxiety and depression, aged between 18 and 50 years. Interventions: Participants were randomly assigned to one of three groups: game-based DTx with RL algorithm (RL algorithm group), game-based DTx without RL algorithm (no algorithm group), and a blank control group. Main Outcomes and Measures: The primary outcomes were reductions in symptoms of anxiety and depression, measured using the Patient Health Questionnaire-9 and Generalized Anxiety Disorder 7-item scales. Response rates and rates of recovery, as well as the impact of demographic variables, were also examined.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 60 years;
2. having a PHQ-9 score or a GAD-7 score upon enrollment;
3. being able to operate a smartphone fluently;
4. having normal vision after correction

Exclusion Criteria:

1. clinical diagnoses of severe psychiatric conditions such as schizophrenia or bipolar disorder;
2. at high risk of suicide or self-harm;
3. having significant cognitive impairments;
4. active substance abuse or dependence;
5. currently undergoing other psychological or pharmacological treatments for depression or anxiety;
6. pregnant individuals or those with postpartum depression, and those with serious physical health conditions that could impact mental health.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
PHQ9 Response | Immeidately after intervention
  A user is said to responded to the intervention if the PHQ9 score dropped no less than 50% compared to the baseline
GAD7 Response | Immeidately after intervention
  A user is said to responded to the intervention if the PHQ9 score dropped no less than 50% compared to the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shao X, Liu L, Zhu X, Tian C, Li D, Zhang L, Liu X, Liu Y, Zhu G, Li L. Personalized game-based digital intervention for relieving depression and anxiety symptoms: a pilot RCT. Npj Ment Health Res. 2025 Jul 3;4(1):27. doi: 10.1038/s44184-025-00141-x. PMID 40610644